CLINICAL TRIAL: NCT05157646
Title: The Relationship Between CFTR Gene Mutations and Exercise Capacity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Student was unable to start the project due to time constraints
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20022243
Record Dates: First submitted 2021-12-01; First posted 2021-12-15 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
Keywords: Exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise trackers (Experimental): Fitbit physical activity trackers
  Interventions: Behavioral: Fitness tracker

INTERVENTIONS:
Behavioral: Fitness tracker — Participants will be asked to wear a Fitbit fitness tracker and report their fitness activity to the study team

SUMMARY:
This study will explore the effect of mutation severity on exercise capacity. Through a better understanding of the association between mutation severity and exercise capacity, clinicians will be more able to predict a given patient's level of independent functioning based on their genes, which is essential information that patients' families want to know upon diagnosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a disease that disrupts the lungs. With an average survival of 40.7 years, this condition affects around 30,000 in the US. Most commonly seen in among those of European descent, CF is present in about 1 in every 2,500 Caucasian newborns. A genetic mutation causes a thick and sticky mucus production in the lungs. Thus, CF patients are more likely to have respiratory failure and lung infections. These symptoms of CF vary among patients and primarily depend on the severity of the gene mutations.Currently, there is not a lot of literature on the relationship between CFTR genes and exercise capacity, highlighting the relevance of this study.

This study is expected to last at least 10 weeks. Participants will be given a Fitbit tracker at the beginning of the study to wear during their participation. Participants are asked to engage in their normal level of physical activity. No one from the research team will have direct access to their Fitbit information. In other words, participants will create an account on the Fitbit website and only participants will be able to see the information on there. A weekly survey about their Fitbit mileage will be given by a research member via phone. The weekly survey will also ask more opinionated questions, regarding any updates on their attitudes toward exercise. At the conclusion of this 10-week study, participants will have the option of keeping their Fitbit tracker. About 50 participants are expected to enroll in this study. At any point of the study, participants will be given the freedom to withdraw their participation.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patient who has been tested positive for a CF mutation of class 1-5.
* Part of the VCU cystic fibrosis program.
* Above 18 years old.

Exclusion Criteria:

* Has not been tested positive for a known CF mutation.
* Not a part of the VCU cystic fibrosis program.
* Cannot be under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in weekly mileage | baseline to 10 weeks
  Participants will report their weekly mileage in a REDCap form

CONTACTS AND LOCATIONS:
Overall Officials: Nauman Chaudary, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No